CLINICAL TRIAL: NCT06638801
Title: Brain Uptrain to Improve Learning and Development: A Randomized Clinical Trial
Brief Title: Brain Uptrain to Improve Learning and Development
Acronym: BUILD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Associate Professor, Neonatologist, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-300013307
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Term Infant; Late Preterm Infant
Keywords: maternal training; cognitive scores; reading; literacy; numeracy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reach Out and Read plus intervention (Experimental): Reach Out and Read Training in addition to coach-led caregiver-implemented early literacy and developmental program
  Interventions: Behavioral: Coach-led caregiver-implemented early literacy and developmental programming; Behavioral: Reach Out and Read Training
- Reach out and Read only (Active Comparator): Reach Out and Read at well child visits
  Interventions: Behavioral: Reach Out and Read Training

INTERVENTIONS:
Behavioral: Coach-led caregiver-implemented early literacy and developmental programming — Caregivers will receive training about child brain development in the first 3 years of life. The training will emphasize the areas of spoken words, physical education, pointer-finger concept, focus and label, reading lessons, and mathematics.
  Arms: Reach Out and Read plus intervention
Behavioral: Reach Out and Read Training — Reach Out and Read parent training

SUMMARY:
The purpose of this study is to see if an early literacy and developmental program in addition to shared reading can increase developmental test scores at 24 months of age. All caregivers of infants in this study will receive shared reading training. Half of the caregivers will be trained in an additional coach-led caregiver-implemented early literacy and numeracy program. Information related to infant development will be collected from parent surveys, medical records, and questionnaires and assessments.

DETAILED DESCRIPTION:
This study will test the hypothesis that in term or late preterm infants who are discharged home from the newborn nursery, a coach-led caregiver-implemented early literacy and developmental program in addition to shared reading, compared with shared reading alone, will increase the Ages and Stages Questionnaire® score at 24 months. This will be a double blind randomized controlled trial with 1:1 parallel allocation using stratified permuted block design. Randomization will be stratified by gestational age (≥ 35 to <38 weeks and ≥ 38 weeks). Randomization of twins and higher orders (when eligible) will be to the same group. Term and late preterm infants ≥ 35 weeks' gestation admitted to the newborn nursery are eligible for inclusion if they are being discharged home. We will exclude infants admitted to the NICU, infants with a known syndrome or major malformation, infants in DHR custody, infants enrolled in a competing study, and infants of families with a primary language other than English or Spanish. All study participants will receive shared reading information at scheduled well-child checks. Caregivers of infants in the intervention group will receive additional coach-led caregiver-implemented early literacy and developmental program. We will complete an ASQ-3 online or by telephone at 12 months, 24 months, and 36 months. We will also measure early literacy at 3 years, 4 years, and 5 years. The primary outcome will be the ASQ-3 scores at 24 months.

ELIGIBILITY:
Inclusion Criteria: inborn at UAB, delivered at more than 35 weeks' gestation, planned for discharge home after initial hospitalization.

-

Exclusion Criteria: a major malformation, a known syndrome, admitted to the NICU, in DHR custody, enrolled in a competing study, and family's primary language is other than English or Spanish.

-

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
ASQ-3 scores | 24 month well-child visit
  The total Ages and Stages Questionnaires 3rd Edition score at 24 months

SECONDARY OUTCOMES:
ASQ-3 scores | 12 month well-child visit
  The total Ages and Stages Questionnaires 3rd Edition score at 12 months
ASQ-3 scores | 36 month well-child visit
  The total Ages and Stages Questionnaires 3rd Edition score at 36 months
ASQ scores below -2SD | 12 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition 2 standard deviations of more below the mean at 12 months
ASQ scores below -2SD | 24 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition 2 standard deviations of more below the mean at 24 months
ASQ scores below -2SD | 36 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition 2 standard deviations of more below the mean at 36 months
ASQ scores below -1SD | 12 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition one standard deviation of more below the mean at 12 months
ASQ scores below -1SD | 24 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition one standard deviation of more below the mean at 24 months
ASQ scores below -1SD | 36 month well-child visit
  The proportion of children with Ages and Stages Questionnaires 3rd Edition one standard deviation of more below the mean at 36 months
Literacy Scores | 36 months
  Get Ready To Read- Revised, McArthur-Bates Communicative Development Inventory, Preschool Language Scales- Fifth Edition scores at 36 months
Literacy Scores | 48 months
  Get Ready To Read- Revised, McArthur-Bates Communicative Development Inventory, Preschool Language Scales- Fifth Edition
Literacy Scores | 60 months
  Get Ready To Read- Revised, McArthur-Bates Communicative Development Inventory, Preschool Language Scales- Fifth Edition scores at 60 months
Kindergarten Readiness | 60 months
  Bracken School Readiness Assessment-Third Edition scores at 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States